CLINICAL TRIAL: NCT03104387
Title: Effects of Diesel Combustion Generated Air Pollution on Cardiovascular Function and Oxidatively Damaged DNA in Healthy Volunteers
Brief Title: Health Effects of Occupational Exposure to Combustion Particles - a Study on Volunteers Performing as Train Conductors
Acronym: BioTrack
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: National Research Centre for the Working Environment, Denmark (Other Government)
Responsible Party: Principal Investigator, Peter Moller, Professor, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: H-16033227; No grant number (Other Grant/Funding Number: Danish Centre for Nanosafety II); 2015-57-0121 case SUND-2016-80 (Other: Danish Data Protection Agency); H-16033227 (Other: Danish Committee on Health Research Ethics for the Capital Region)
Record Dates: First submitted 2017-03-23; First posted 2017-04-07 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Cardiovascular Function; Genotoxicity
Keywords: Air pollution; Diesel exhaust; Ultrafine particles; Vascular function; Endothelium function; Heart rate variability; DNA damage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diesel train - exposure scenario (Experimental): The same study person will be exposed to two different scenarios, at different times and for three consecutive days. It will be a lag time of 2 weeks between each exposure scenario. The "exposure" scenario is defined as a workday (6 hours) on the diesel ME-driven model regional train. The Diesel Train Scenario is performed twice. After the scenario completion (on the third day in defined train routes) the vascular function, lung function, blood and urine samplings are performed.
  Interventions: Other: Diesel train
- Electric train - low exposure scenario (Sham Comparator): The same study person will be exposed to two different scenarios, at different times and for three consecutive days. It will be a lag time of 2 weeks between each exposure scenario. The "low exposure" scenario is defined as a workday (6 hours) on the electric train. The Diesel Train Scenario is performed twice. After the scenario completion (on the third day in defined train routes) the vascular function, lung function, blood and urine samplings are performed.
  Interventions: Other: Electric train

INTERVENTIONS:
Other: Electric train — Exposure to air with low level of ultrafine particles (Electric train)
  Arms: Electric train - low exposure scenario
Other: Diesel train — Exposure to air with high level of ultrafine particles (Diesel train)
  Arms: Diesel train - exposure scenario

SUMMARY:
Ambient air pollution is a complex mixture of gaseous pollutants and particulate matter (PM). PM has a recognized important role in human health. There is a strong scientific consensus on the independent association of PM and adverse cardiovascular and respiratory effects, as well as cancer. It is reasonable to expect that the smaller particles (ultrafine particles, UFP) may have an enhanced toxicity relative to other PM size fractions, due to physical properties and potential to translocation beyond the lung.

A recent Danish report concluded that train conductors on a working day, and in two specific diesel engine trains, are exposed to higher concentrations of diesel exhaust than by constant stay in a busy street. Indeed, the average exposure for train conductors on such engines was around 100,000-150,000 UFP per cm3 as compared with around 40,000 per cm3 on a busy street in Copenhagen [1]. The aim of this study is to investigate if this occupational exposure is associated with vascular and respiratory impairment and DNA damage.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Legally competent subjects

Exclusion Criteria:

* Current smokers
* Pregnancy
* Alcohol and drug abuse
* Prescriptionary use of anti-inflammatory or cardiovascular medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Reactive hyperemia index measured by peripheral arterial tonometry | Peripheral arterial tonometry is assessed after each exposure scenario (on the third day after 6 hours on defined train routes per day)
  The primary outcome will be measured in the form of post-ischemic variation followed by the measurement of the vasomotor function after the administration of nitroglycerin, to allow the investigation of the endothelium independent vasodilatation. The portable device EndoPAT 2000 will be used (Itamar Medical Ltd, Israel) [2-6].
Heart rate variability | Assessed after each exposure scenario (on the third day after 6 hours on defined train routes per day)
  Heart rate variability is measured with the EndoPAT 2000 device during baseline recording. It includes time domain measures (SDNN, pNN50 and RMSSD), high (HF) and low frequency (LF) components as well as LF/HF ratio, based on measurements over 5 minutes.
DNA damage in peripheral blood mononuclear cells | Blood is sampled, prepared and stored after each exposure scenario (on the third day after 6 hours on defined train routes per day). Analysis is performed after sample collection completion.
  The levels of strand breaks and formamidopyrimidine-DNA-glycosylase (FPG) sites are measured with the single cell gel electrophoresis assay (comet assay) [7-13]

SECONDARY OUTCOMES:
Lung function | The lung function is assessed after each exposure scenario (on the third day after 6 hours on defined train routes per day)
  The lung function is measured with EasyOne 2001 spirometer device (Switzerland). Lung function measurements includes forced vital capacity (FVC), forced expiratory volume after 1 second (FEV1), peak expiratory flow (PEF) and FEV1/FVC.
Systemic inflammatory markers | Blood is sampled, prepared and stored after each exposure scenario (on the third day after 6 hours on defined train routes per day). Analysis is performed after sample collection completion.
  Acute phase reactants, pro-inflammatory cytokines and cell adhesion molecules
Urinary excretion of 1-hydroxypyrene | Morning urine is sampled, prepared and stored after each exposure scenario (on the morning of the third day after two days with 6 hours on defined train routes). Analysis is performed after sample collection completion.
  The urinary biomarker of exposure to polycyclic aromatic hydrocarbons, 1-hydroxypyrene, is measured with reverse-phase HPLC and standardized for diuresis with the concentration of creatinine
Serum/plasma bioactivity | Blood is sampled, prepared and serum is stored after each exposure scenario (on the third day after 6 hours on defined train routes per day). Analysis is performed after sample collection completion.
  To assess the potential effects on vascular and endothelial function [14, 15]

OTHER OUTCOMES:
Augmentation index | Assessed after each exposure scenario (on the third day after 6 hours on defined train routes per day)
  Measured with the EndoPAT 2000 device during baseline recording.
Blood pressure | Assessed after each exposure scenario (on the third day after 6 hours on defined train routes per day)
  Measured with an aneroid sphygmomanometer.
Heart rate | Assessed after each exposure scenario (on the third day after 6 hours on defined train routes per day)
  Measured with the EndoPAT 2000 device during baseline recording.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Moller, PhD, Principal Investigator — University of Copenhagen
Locations (1):
- University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karottki G, Loft S. Rapport vedroerende maaling af udsaettelse for ultrafine partikler blandt ansatte i DSB, 1-48, 2015.
- [Result] Brauner EV, Forchhammer L, Moller P, Barregard L, Gunnarsen L, Afshari A, Wahlin P, Glasius M, Dragsted LO, Basu S, Raaschou-Nielsen O, Loft S. Indoor particles affect vascular function in the aged: an air filtration-based intervention study. Am J Respir Crit Care Med. 2008 Feb 15;177(4):419-25. doi: 10.1164/rccm.200704-632OC. Epub 2007 Oct 11. PMID 17932377
- [Result] Olsen Y, Karottki DG, Jensen DM, Beko G, Kjeldsen BU, Clausen G, Hersoug LG, Holst GJ, Wierzbicka A, Sigsgaard T, Linneberg A, Moller P, Loft S. Vascular and lung function related to ultrafine and fine particles exposure assessed by personal and indoor monitoring: a cross-sectional study. Environ Health. 2014 Dec 15;13:112. doi: 10.1186/1476-069X-13-112. PMID 25512042
- [Result] Karottki DG, Spilak M, Frederiksen M, Gunnarsen L, Brauner EV, Kolarik B, Andersen ZJ, Sigsgaard T, Barregard L, Strandberg B, Sallsten G, Moller P, Loft S. An indoor air filtration study in homes of elderly: cardiovascular and respiratory effects of exposure to particulate matter. Environ Health. 2013 Dec 28;12:116. doi: 10.1186/1476-069X-12-116. PMID 24373585
- [Result] Hemmingsen JG, Rissler J, Lykkesfeldt J, Sallsten G, Kristiansen J, Moller P P, Loft S. Controlled exposure to particulate matter from urban street air is associated with decreased vasodilation and heart rate variability in overweight and older adults. Part Fibre Toxicol. 2015 Mar 19;12:6. doi: 10.1186/s12989-015-0081-9. PMID 25890359
- [Result] Brauner EV, Moller P, Barregard L, Dragsted LO, Glasius M, Wahlin P, Vinzents P, Raaschou-Nielsen O, Loft S. Exposure to ambient concentrations of particulate air pollution does not influence vascular function or inflammatory pathways in young healthy individuals. Part Fibre Toxicol. 2008 Oct 6;5:13. doi: 10.1186/1743-8977-5-13. PMID 18837984
- [Result] Forchhammer L, Moller P, Riddervold IS, Bonlokke J, Massling A, Sigsgaard T, Loft S. Controlled human wood smoke exposure: oxidative stress, inflammation and microvascular function. Part Fibre Toxicol. 2012 Mar 27;9:7. doi: 10.1186/1743-8977-9-7. PMID 22452928
- [Result] Brauner EV, Forchhammer L, Moller P, Simonsen J, Glasius M, Wahlin P, Raaschou-Nielsen O, Loft S. Exposure to ultrafine particles from ambient air and oxidative stress-induced DNA damage. Environ Health Perspect. 2007 Aug;115(8):1177-82. doi: 10.1289/ehp.9984. PMID 17687444
- [Result] Danielsen PH, Brauner EV, Barregard L, Sallsten G, Wallin M, Olinski R, Rozalski R, Moller P, Loft S. Oxidatively damaged DNA and its repair after experimental exposure to wood smoke in healthy humans. Mutat Res. 2008 Jul 3;642(1-2):37-42. doi: 10.1016/j.mrfmmm.2008.04.001. Epub 2008 Apr 14. PMID 18495177
- [Result] Hemmingsen JG, Jantzen K, Moller P, Loft S. No oxidative stress or DNA damage in peripheral blood mononuclear cells after exposure to particles from urban street air in overweight elderly. Mutagenesis. 2015 Sep;30(5):635-42. doi: 10.1093/mutage/gev027. Epub 2015 Apr 22. PMID 25904586
- [Result] Moller P, Danielsen PH, Karottki DG, Jantzen K, Roursgaard M, Klingberg H, Jensen DM, Christophersen DV, Hemmingsen JG, Cao Y, Loft S. Oxidative stress and inflammation generated DNA damage by exposure to air pollution particles. Mutat Res Rev Mutat Res. 2014 Oct-Dec;762:133-66. doi: 10.1016/j.mrrev.2014.09.001. Epub 2014 Sep 16. PMID 25475422
- [Result] Moller P, Hemmingsen JG, Jensen DM, Danielsen PH, Karottki DG, Jantzen K, Roursgaard M, Cao Y, Kermanizadeh A, Klingberg H, Christophersen DV, Hersoug LG, Loft S. Applications of the comet assay in particle toxicology: air pollution and engineered nanomaterials exposure. Mutagenesis. 2015 Jan;30(1):67-83. doi: 10.1093/mutage/geu035. PMID 25527730
- [Result] Moller P, Loft S. Oxidative damage to DNA and lipids as biomarkers of exposure to air pollution. Environ Health Perspect. 2010 Aug;118(8):1126-36. doi: 10.1289/ehp.0901725. Epub 2010 Apr 27. PMID 20423813
- [Result] Aragon M, Erdely A, Bishop L, Salmen R, Weaver J, Liu J, Hall P, Eye T, Kodali V, Zeidler-Erdely P, Stafflinger JE, Ottens AK, Campen MJ. MMP-9-Dependent Serum-Borne Bioactivity Caused by Multiwalled Carbon Nanotube Exposure Induces Vascular Dysfunction via the CD36 Scavenger Receptor. Toxicol Sci. 2016 Apr;150(2):488-98. doi: 10.1093/toxsci/kfw015. Epub 2016 Jan 21. PMID 26801584
- [Result] Aragon MJ, Chrobak I, Brower J, Roldan L, Fredenburgh LE, McDonald JD, Campen MJ. Inflammatory and Vasoactive Effects of Serum Following Inhalation of Varied Complex Mixtures. Cardiovasc Toxicol. 2016 Apr;16(2):163-71. doi: 10.1007/s12012-015-9325-z. PMID 25900702
- [Derived] Andersen MHG, Frederiksen M, Saber AT, Wils RS, Fonseca AS, Koponen IK, Johannesson S, Roursgaard M, Loft S, Moller P, Vogel U. Health effects of exposure to diesel exhaust in diesel-powered trains. Part Fibre Toxicol. 2019 Jun 11;16(1):21. doi: 10.1186/s12989-019-0306-4. PMID 31182122